CLINICAL TRIAL: NCT06815471
Title: Corticotrophin Releasing Factor 2 for the Treatment of Worsening Heart Failure (WHF) - The CRAFT-WHF Study
Brief Title: CRF2 Agonist for the Treatment of Worsening Heart Failure
Acronym: CRAFT-WHF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Corteria Pharmaceuticals (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COR1167-201
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Worsening Heart Failure
Keywords: COR-1167; Hospitalised heart failure; WHF

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor CRO
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- COR-1167 low dose (Experimental)
  Interventions: Drug: COR-1167
- COR-1167 intermediate dose (Experimental)
  Interventions: Drug: COR-1167
- COR-1167 high dose (Experimental)
  Interventions: Drug: COR-1167
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COR-1167 — 28-day treatment
  Arms: COR-1167 high dose; COR-1167 intermediate dose; COR-1167 low dose
Drug: Placebo — 28-day treatment
  Arms: Placebo

SUMMARY:
This study assesses the effects of the investigational drug COR-1167 in subjects hospitalised due to worsening of heart failure (HF)

DETAILED DESCRIPTION:
This is a phase 2b, randomized, double-blind, placebo-controlled study designed to assess the dose-dependent effects of 3 doses of the corticotropin-releasing factor type 2 (CRF2) peptide agonist, COR-1167, in subjects with WHF, defined as subjects requiring urgent administration of intravenous (i.v.) diuretics due to worsening of signs and symptoms of heart failure (HF) associated with volume overload

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Heart failure hospitalization (HFH) during previous 12 months
* Prescribed an oral loop diuretic for at least 1 month preceding the index event
* NT-proBNP ≥1,000 pg/mL or BNP ≥250 pg/mL
* Requires treatment with i.v. diuretics for volume overload
* At least 1 risk factor for diuretic resistance
* Admitted to the hospital not more than 48 hours prior to randomization

Exclusion Criteria:

* Index event primarily triggered by an acute event (e.g. AMI, PE, arrhythmia)
* Requirement for i.v. inotropic therapy or i.v. vasodilators, mechanical ventilation, high-flow oxygen therapy, or NIV
* Requirement for, or planned use of LVADs, IABP, or any type of MCS
* History of solid organ transplant or active on a transplant list
* SBP <100 mmHg
* eGFR < 20 mL/min/1.73 m2
* CABG, PCI, implantation of CRT, heart valve procedure or any cardiac surgery within 1 month prior to screening or planned during the study
* Severe stenotic cardiac valvular disease
* Severe chronic pulmonary disease requiring chronic steroid therapy or chronic oxygen therapy (> 2 L/min)
* Uncorrected severe hyperthyroidism or hypothyroidism
* Severe restrictive, obstructive, or infiltrative cardiomyopathy
* Body weight < 70 kg
* Use of any investigational drug(s) within 5 half-lives of screening
* At high risk of death (defined as life expectancy ≤1 year) from causes other than heart failure or any disease that, in the opinion of the Investigator, will preclude their safe participation in this study, and will make implementation of the protocol or interpretation of the study results difficult
* Presence of any other conditions (e.g. geographic, social) actual or anticipated, that the Investigator feels would restrict or limit the subject's participation or compliance with all study procedures Subject is the Investigator or any Subinvestigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Natriuresis | 24 hours
  Urinary sodium excretion
Body weight | 7 days
  Changes in body weight
NT-proBNP | 7 days
  Changes in NT-proBNP
Kansas City Cardiomyopathy Questionnaire (KCCQ)-Total Symptom Score (TSS) | 28 days
  Changes in KCCQ-TSS - The score ranges from 0 to 100 with higher score indicating a better health status
Left Atrial Volume index (LAVi) | 2 days
  Changes in LAVi - LAV-i is an index of cardiac function measured by echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, MD, Study Chair — Yale University
Locations (43):
- United States (5):
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Cone Health Moses Cone Hospital, Greensboro, North Carolina
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - Ohio State University, Columbus, Ohio
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
- Czechia (3):
  - Fakultní nemocnice Ostrava, Ostrava, Czech Republic
  - Sdružené zdravotnické zařízení Krnov, Krnov
  - Nemocnice Slaný, Slaný
- Georgia (9):
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - LTD "Israeli-Georgian Medical Research Clinic Healthycore", Tbilisi
  - Acad. G. Chapidze Emergency Cardiology Center LTD, Department of Internal Medicine and Medical Research, Tbilisi
  - Acad. G.Chapidze Emergency Cardiology Center, LTD, Department of Multi-center Clinical Trials, Tbilisi
  - Bokhua Memorial Cardiovascular Center LTD, Tbilisi
  - St. Michael's Hospital LLC, Tbilisi
  - Tbilisi Heart and Vascular Clinic, LTD, Tbilisi
  - Georgian Dutch Hospital, Tbilisi
  - LTD Tbilisi Heart Center, Tbilisi
- Hungary (5):
  - Semmelweis Egyetem, Általános Orvostudományi Kar, Városmajori Szív- és Érgyógyászati Klinika, Budapest
  - Budapesti Uzsoki Utcai Kórház, Kardiológia Osztály, Budapest
  - Pécsi Tudományegyetem, Klinikai Központ, I. sz. Belgyógyászati Klinika, Pécs
  - Szegedi Tudományegyetem, Általános Orvostudományi Kar, Családorvosi Intézet, Szeged
  - Zala Vármegyei Szent Rafael Kórház, Kardiológiai Osztály, Zalaegerszeg
- Poland (5):
  - Klinika Kardiologii i Chorób Wewnętrznych z Oddziałem Intensywnego Nadzoru Kardiologicznego (OINK), Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Zespół Opieki Zdrowotnej w Klodzku, Oddzial Kardiologii, Kłodzko
  - Kliniczny Szpital Wojewódzki nr 2 im. Św. Jadwigi Królowej w Rzeszowie, Rzeszów
  - Oddział Kliniczny Kardiologii i Intensywnej Terapii Kardiologicznej, Torun
  - Instytut Chorób Serca, Zakład Badań Klinicznych Chorób Układu Krążenia, Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw
- Romania (3):
  - Emergency County Clinical Hospital Arad, Cardiology department, Arad
  - Craiova County Emergency Clinical Hospital, Craiova
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- Serbia (8):
  - Clinical Hospital Center "Dr Dragisa Misovic Dedinje", Belgrade
  - Institute for Cardiovascular Diseases Dedinje, Belgrade
  - University Clinical Center of Serbia, Clinic for Cardiology, Department for the testing and treatment of congenital and acquired heart defects, Belgrade
  - University Clinical Center of Serbia, Clinic for Cardiology, Emergency Cardiology Department, Belgrade
  - University Clinical Center of Serbia, Clinic for Cardiology, Heart Failure Ward, Belgrade
  - University Clinical Center Kragujevac, Clinic for Cardiology, Kragujevac
  - General Hospital Leskovac, Cardiology Department, Leskovac
  - University Clinical Center Nis, Clinic for Cardiology, Niš
- Spain (5):
  - Hospital Universitario Ramon y Cajal, Fuencarral-El Pardo, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Hospital Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No
This is not a phase 3 trial that would benefit from IPD sharing

REFERENCES:
- [Result] Rademaker MT, Charles CJ, Ellmers LJ, Lewis LK, Nicholls MG, Richards AM. Prolonged urocortin 2 administration in experimental heart failure: sustained hemodynamic, endocrine, and renal effects. Hypertension. 2011 Jun;57(6):1136-44. doi: 10.1161/HYPERTENSIONAHA.111.173203. Epub 2011 May 2. PMID 21536988
- [Result] Rademaker MT, Charles CJ, Nicholls MG, Richards AM. Urocortin 2 inhibits furosemide-induced activation of renin and enhances renal function and diuretic responsiveness in experimental heart failure. Circ Heart Fail. 2009 Nov;2(6):532-40. doi: 10.1161/CIRCHEARTFAILURE.109.861336. Epub 2009 Sep 22. PMID 19919977
- [Result] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Result] Chan WY, Frampton CM, Crozier IG, Troughton RW, Richards AM. Urocortin-2 infusion in acute decompensated heart failure: findings from the UNICORN study (urocortin-2 in the treatment of acute heart failure as an adjunct over conventional therapy). JACC Heart Fail. 2013 Oct;1(5):433-41. doi: 10.1016/j.jchf.2013.07.003. Epub 2013 Sep 11. PMID 24621976
- [Result] Rubio-Gracia J, Demissei BG, Ter Maaten JM, Cleland JG, O'Connor CM, Metra M, Ponikowski P, Teerlink JR, Cotter G, Davison BA, Givertz MM, Bloomfield DM, Dittrich H, Damman K, Perez-Calvo JI, Voors AA. Prevalence, predictors and clinical outcome of residual congestion in acute decompensated heart failure. Int J Cardiol. 2018 May 1;258:185-191. doi: 10.1016/j.ijcard.2018.01.067. PMID 29544928
- [Result] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):399-410. doi: 10.1161/01.cir.0000442015.53336.12. No abstract available. PMID 24446411